CLINICAL TRIAL: NCT06513000
Title: Evaluation Of Dry Eye After Uneventful Phacoemulsification
Brief Title: Dryness Difference Between Before and After Phacoemulsification
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Samir, Doctor, Sohag University
Other Study IDs: Dryness post phaco
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dry eye diagnostic system — following tests:
  1. Non-invasive tear film break up time (TBUT), a parameter of tear film stability.
  2. Non-invasive tear meniscus height.
  3. Evaluation of Meibomian glands function.
  4. Lipid layer thickness.
  5. Eyelid margin.
  6. Analysis of conjunctival hyperemia.
  7. Cornea sodium fluorescein staining.
  8. Schirmer I test

SUMMARY:
The aim of this study is to compare tear film and tear film secretion before and after phacoemulsificaton cataract surgery

DETAILED DESCRIPTION:
The tear film is a thin fluid layer overlies the ocular surface and provides the interface between the ocular surface and the external environment.

* It consists of three layers (lipid, aqueous and mucous) which act together to protect the corneal and conjunctival tissues and keeping them healthy.
* The superficial lipid layer is secreted by meibomian glands and functions as a smooth optical surface, reduces surface tension of the tear film, prevents anterior migration of aqueous tears on to the lid margin and retards evaporation .
* The Mucous layer is secreted by the goblet cells of the conjunctiva. It contains mucins that is very essential for lubrication, and wetting.
* The aqueous tear layer is mainly produced by the main lacrimal glands with small amounts produced by the goblet cells in the conjunctiva and accessory lacrimal glands and This layer acts by providing oxygen and nutrients to the avascular corneal tissue, washing away tissue debris, toxins, and foreign bodies, and also protecting the ocular surface from microbes.
* Cataract is the common cause of vision loss in the developing countries, also its rate of incidence increases with aging. So it is essential for those patients to undergo cataract surgeries to improve their vision and protect them from blindness.
* Phacoemulsification is the most recent cataract surgery at which a small incision is done then the ultrasonic power is used to fragment and emulsify the cataract. It was first introduced by Dr. Charlies Kelman and now Most surgeons prefer phacoemulsification surgery because of less postoperative astigmatism, faster stabilization of vision and refraction, and less postoperative inflammation
* Some surgical interventions related to the anterior segment may also cause dry eye and aggravate the symptoms of pre-existing dry eye, like PRK, LASIK, and cataract surgery by extra capsular cataract extraction, because a large incision is created in the eye during the procedure that sometimes damages the cornea and also can occur with phacoemulsification with a smaller incision.
* There are many tests that are used to estimate the degree of dryness and its severity which measure tear stability, tear production, and the presence of ocular surface disorders like Schirmer's test , which is used to evaluate tear production and the severity of dry eye by estimating the amount of special filter paper wetting that is put in the lower fornix for 5 minutes, and the Tears Break Up Time test, which is important to evaluate the tear film stability and evaporation.
* In this study we aim to evaluate dry eye affection after phacoemulsification whether it is worsen or not and the degree of increased dryness especially that dry eye syndrome is very common in our community and how phacoemulsification is now a frequent and preferred operation.

After taking a good detailed history The following assessments were performed in each patient before surgery and at the 2-week and 1-, 3-, and 6-month follow-up visits by the following tests:

1. Non-invasive tear film break up time (TBUT), a parameter of tear film stability.
2. Non-invasive tear meniscus height.
3. Evaluation of Meibomian glands function.
4. Lipid layer thickness.
5. Eyelid margin.
6. Analysis of conjunctival hyperemia.
7. Cornea sodium fluorescein staining.

   * Schirmer I test, a measure of basic and reflex tear secretion, was performed without anesthesia. This test was performed by placing Schirmer strips over the lower lid margin; the strip wetting was measured and recorded in millimeters.
   * Dry eye symptoms patients were classified as having dry eye disease if they reported experiencing one or more of the primary symptoms (soreness, scratchiness, dryness, grittiness, burning) often or constantly, the TBUT value was less than 10 seconds, and in Schirmer test I there is less than 10 mm wetting of filter paper for a period of 6 months or more after surgery.
   * Visual acuity before and after surgery.
   * Anterior segment examination by slit lamp.

ELIGIBILITY:
Inclusion criteria:

* Cataract patients.
* Cases within age > 45 years old.

Exclusion criteria:

* Patients with ocular surface diseases and eyelid abnormality.
* Patients receive ocular or systemic medications, that interfere with tear film production and stability (e.g. topical eye drops that contain preservatives, antihistaminic drugs, anticholinergic drugs, contraceptive pills).
* Patients with systemic diseases like diabetes, HTN, rheumatoid arthritis. - Patients underwent previous ocular surgeries that interfere with tears instability or production (e.g. refractive surgery, keratoplasty, eyelid surgeries, pterygium excision).
* Patients with a history of trauma, chemical burn, overusing contact lens (due to damaging the conjunctiva and the goblet cells, also corneal sensitivity reduction).

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: this study included 100 cataract patients, with age above 45 years old who underwent uncomplicated phacoemulsification surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation Of Dryness Post Phacoemulcification In Non Complicated Cases using tear film break up time in seconds. | Before the operation and 2-week and 1, 3, and 6 month after the operation
  Analysis of dryness before and after uncomplicated phacoemulsification using tear film break up time in seconds.
Evaluation Of Dryness Post Phacoemulcification In Non Complicated Cases using tear meniscus height in millimeters. | Before the operation and 2-week and 1, 3, and 6 month after the operation
  Analysis of dryness before and after uncomplicated phacoemulsification using tear meniscus height in millimeters.
Evaluation Of Dryness Post Phacoemulcification In Non Complicated Cases using Lipid layer thickness in nanometers. | Before the operation and 2-week and 1, 3, and 6 month after the operation
  Analysis of dryness before and after uncomplicated phacoemulsification using Lipid layer thickness in nanometers..

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Gamal eldeen, Professor, Study Director — Sohag University; Mahmoud Mohamed farouk, Professor, Study Chair — Sohag University; Hany Mahmoud, Lecturer, Study Chair — Sohag University; Mohamed samir zayed, resident, Principal Investigator — Tahta ophthalmology hospital
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Background] Qin Y, Pan ZQ. [Recent advances in dry eye: etiology, pathogenesis and management]. Zhonghua Yan Ke Za Zhi. 2013 Sep;49(9):857-63. Chinese. PMID 24330938
- [Background] Moss SE, Klein R, Klein BE. Long-term incidence of dry eye in an older population. Optom Vis Sci. 2008 Aug;85(8):668-74. doi: 10.1097/OPX.0b013e318181a947. PMID 18677233
- [Background] Mertzanis P, Abetz L, Rajagopalan K, Espindle D, Chalmers R, Snyder C, Caffery B, Edrington T, Simpson T, Nelson JD, Begley C. The relative burden of dry eye in patients' lives: comparisons to a U.S. normative sample. Invest Ophthalmol Vis Sci. 2005 Jan;46(1):46-50. doi: 10.1167/iovs.03-0915. PMID 15623753
- [Background] Pflugfelder SC, Stern ME. Biological functions of tear film. Exp Eye Res. 2020 Aug;197:108115. doi: 10.1016/j.exer.2020.108115. Epub 2020 Jun 16. PMID 32561483
- [Background] Xue W, Zhu MM, Zhu BJ, Huang JN, Sun Q, Miao YY, Zou HD. Long-term impact of dry eye symptoms on vision-related quality of life after phacoemulsification surgery. Int Ophthalmol. 2019 Feb;39(2):419-429. doi: 10.1007/s10792-018-0828-z. Epub 2018 Feb 1. PMID 29392638